CLINICAL TRIAL: NCT02906605
Title: An Open-label, Randomized, Phase 2 Study of the Clinical Activity and Safety of JNJ-64041809, a Live Attenuated Listeria Monocytogenes Immunotherapy, in Combination With Apalutamide Versus Apalutamide in Subjects With Metastatic Castration-resistant Prostate Cancer
Brief Title: A Study of the Clinical Activity and Safety of JNJ-64041809, a Live Attenuated Listeria Monocytogenes Immunotherapy, in Combination With Apalutamide Versus Apalutamide in Subjects With Metastatic Castration-resistant Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study start delayed due to pending collection and analysis of additional phase 1 data.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108224; 64041809PCR2002 (Other: Janssen Research & Development, LLC); 2016-001917-26 (EudraCT Number)
Record Dates: First submitted 2016-09-15; First posted 2016-09-20 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Prostatic Neoplasms, Castration-Resistant
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant | interventions — apalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- JNJ-809 plus Apalutamide (Group A) (Experimental): JNJ-809 given as an infusion and Apalutamide 240 milligram (mg) daily.
  Interventions: Drug: JNJ-809; Drug: Apalutamide
- Apalutamide (Group B) (Experimental): Apalutamide 240 mg orally daily.
  Interventions: Drug: Apalutamide

INTERVENTIONS:
Drug: JNJ-809 — JNJ-809 (1*10^9) colony forming units (CFU) given as an infusion.
  Arms: JNJ-809 plus Apalutamide (Group A)
Drug: Apalutamide — Apalutamide 240 mg orally daily.

SUMMARY:
The purpose of this study is to evaluate if the anti-tumor activity of JNJ-809 combined with apalutamide is improved compared with apalutamide alone for subjects with metastatic castration-resistant prostate cancer (mCRPC).

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the prostate
* Metastatic disease as documented by technetium-99m (99mTc) bone scan or metastatic lesions by computed tomography (CT) or magnetic resonance imaging (MRI) scans
* Surgically or medically castrated, with testosterone levels of less than (<)50 nanogram per deciliter (ng/dL)
* Castration-resistant prostate cancer documented by time to prostate-specific antigen (PSA) increase during continuous treatment with androgen deprivation therapy (ADT) OR radiographic progression of soft tissues OR radiographic progression of bone according to PCWG3

Exclusion Criteria:

* Predominately small cell or neuroendocrine carcinoma of the prostate
* Known brain metastases (even if treated) or untreated epidural spread
* Prior chemotherapy for prostate cancer, except if administered in the adjuvant/neoadjuvant setting, or up to 6 cycles of docetaxel for metastatic hormone-sensitive prostate cancer
* Treatment with medications known to lower the seizure threshold or any investigational agent that were not discontinued or substituted greater than or equal to (>=)28 days prior to randomization

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Time to Prostate-specific Antigen (PSA) Progression | approximately 2 years
  Time to PSA progression will be measured using Prostate Cancer Working Group 3 (PCWG3).

SECONDARY OUTCOMES:
PSA Doubling Time (PSADT) | approximately 2 years
  The PSADT will be determined using the method as recommended by PCWG3 criteria.
Radiographic Progression-free Survival | approximately 2 years
  Radiographic progression-free survival, is defined as the time from the date of randomization to the date of radiographic progression or death, whichever occurs first.
Time to Unequivocal Clinical Progression | approximately 2 years
  Time to unequivocal clinical progression defined as the time from the date of randomization to the date of unequivocal clinical progression as evaluated by the investigator.
Overall Survival | approximately 2 years
  Overall survival defined as time from the date of randomization to death from any cause.
Number of Participants With Adverse Events (AEs) as a Measure of Safety and Tolerability | approximately 2 years
  Comparison of the AE profiles of the two treatment groups.
Blood Culture and Shedding Profile of JNJ-809 From Cultured Samples of Feces, Urine, and Saliva | approximately 2 years
  Blood culture samples will be collected after the mandatory prophylactic antibiotic therapy. Bacterial shedding will be evaluated from cultured samples of feces by stool or rectal swab, urine, and sputum.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- New York, New York, United States